CLINICAL TRIAL: NCT02296177
Title: Evidence Based Dissemination for Mammography Adherence in Safety Net Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linda Highfield, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-14-0269
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: evidence-based intervention; mammography; underserved population
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control group will receive the standard practice of care related to mammography phone call reminders. If a clinic currently conducts reminders, they will receive that standard call. If no reminders are done, then they will not receive a call during the control period.
- Intervention (Active Comparator): The intervention group will receive a reminder call about their upcoming appointment that assesses their intent to attend the appointment and counsels them through barriers to attendance. The call is conducted by a trained patient navigator using an adapted NCI RTIP to increase mammography appointment adherence.
  Interventions: Behavioral: Peace of Mind Program

INTERVENTIONS:
Behavioral: Peace of Mind Program — The Peace of Mind Program (PMP) is a telephone counseling program based on the Transtheoretical Model of Change, with messages matched to readiness (assessed with a stage of change question)and barriers identified by women who are non-adherent to mammography. The program telephone protocol guides counselors to assess a woman's readiness to be screened and counsel her through barriers to increase appointment keeping.
  Arms: Intervention

SUMMARY:
Breast cancer is the most common cancer and the second leading cause of cancer related death in American women. Regular screening, early diagnosis, and timely treatment initiation have been shown to reduce breast cancer morbidity and mortality. However, disparities continue to exist across the breast cancer continuum for underserved women, particularly minority women. The reduction of disparities in breast cancer outcomes is a major goal of Healthy People 2020 and the National Cancer Institute. However, the preventable burden of late stage breast cancer will continue until the investigators close the gap between what is known about prevention and what is implemented in the community. Although many sources of information exist about theory and [theory-] and evidence-based interventions (EBIs) to promote mammography screening, their adoption and use in the community has been limited and haphazard at best.

DETAILED DESCRIPTION:
In order to effectively reach underserved women and reduce breast cancer disparities, D&I efforts should target the healthcare delivery system where these women receive service - the so called "safety net". Within the safety net, federally qualified health centers (FQHCs), provide comprehensive primary health care services for underserved communities regardless of ability to pay, including mammography screening. Our team has successfully pilot tested a National Cancer Institute research tested intervention program (RTIP) with underserved women and were able to reduce no-show rates from 44% to 19%. In order to accelerate the adoption and implementation of our EBI within the safety net, the investigators will use a two-step approach based on the consolidated framework for implementation research (CFIR), and intervention mapping. The investigators will actively disseminate the EBI through a unique breast health collaborative with a wide membership of FQHCs, support implementation through training and evaluate the adoption, implementation, sustainment and effectiveness of the EBI. The investigators will use a clinic clustered stepped wedge design for implementation in FQHCs.

ELIGIBILITY:
Inclusion Criteria:

* Underserved as defined by income <=200% of the federal poverty level for a family of four
* Uninsured
* In need of mammography screening; has received clinical breast exam and referral to screening
* Has upcoming screening appointment

Exclusion Criteria:

-

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4448 (Actual)
Dates: Start 2015-07; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Mammography Appointment Adherence | 12 months
  Appointment attendance will be taken from the electronic health record for both control and intervention patients

SECONDARY OUTCOMES:
Cancellations or rescheduled appointments | 12 months
  Patients who cancelled and rescheduled will be taken from the electronic health record for both control and intervention patients

CONTACTS AND LOCATIONS:
Overall Officials: Linda Highfield, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holcomb J, Rajan SS, Ferguson GM, Sun J, Walton GH, Highfield L. Implementation of an Evidence-Based Intervention with Safety Net Clinics to Improve Mammography Appointment Adherence Among Underserved Women. J Cancer Educ. 2023 Feb;38(1):309-318. doi: 10.1007/s13187-021-02116-w. Epub 2021 Nov 25. PMID 34822118
- [Derived] Highfield L, Valerio MA, Fernandez ME, Eldridge-Bartholomew LK. Development of an Implementation Intervention Using Intervention Mapping to Increase Mammography Among Low Income Women. Front Public Health. 2018 Oct 26;6:300. doi: 10.3389/fpubh.2018.00300. eCollection 2018. PMID 30416992
- [Derived] Highfield L, Rajan SS, Valerio MA, Walton G, Fernandez ME, Bartholomew LK. A non-randomized controlled stepped wedge trial to evaluate the effectiveness of a multi-level mammography intervention in improving appointment adherence in underserved women. Implement Sci. 2015 Oct 14;10:143. doi: 10.1186/s13012-015-0334-x. PMID 26464110